CLINICAL TRIAL: NCT07146659
Title: Comparison of Operative Hysteroscopy Performed in the Operating Room Versus Outpatient Settings : A Prospective Observational Study
Brief Title: Comparison of Operative Hysteroscopy Performed in the Operating Room Versus Outpatient Settings
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: HOPE
Record Dates: First submitted 2025-07-18; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-07

CONDITIONS: Fibroid Uterus; Polyp Uterus; Retained Products of Conception
Keywords: Hysteroscopy; Operative hysteroscopy; Outpatient ambulatory; Patient satisfaction; Outpatient hysteroscopy; Complications
MeSH Terms: conditions — Leiomyoma; Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Operative hysteroscopy in the operating room: Operative hysteroscopy in the operating room: Procedures performed under general or regional anesthesia in a surgical setting (either ambulatory or conventional hospitalization).
- Operative hysteroscopy in the outpatient setting: Operative hysteroscopy in the outpatient setting: Procedures performed in a consultation room without general or regional anesthesia, using local anesthesia if needed

SUMMARY:
This is an observational prospective monocentric study which aims to compare operative hysteroscopies performed in the operating room under general or loco-regional anesthesia and those performed outside the operating room (outpatient operative hysteroscopy). The primary outcome is the success rate of the procedure. Secondary outcomes include postoperative pain, patient satisfaction, complications, and time to return to work.

DETAILED DESCRIPTION:
Operative hysteroscopy is a key technique for the treatment of intrauterine pathologies such as endometrial polyps, submucosal fibroids, retained products of conception. Traditionally, operative hysteroscopies are performed in the operating room under general or regional anesthesia, requiring either ambulatory or inpatient hospitalization.

In recent years, advances in hysteroscopic instrumentation and procedural techniques have made it possible to perform selected operative hysteroscopies in outpatient settings (consultation office) without general or regional anesthesia. Several studies have demonstrated the feasibility, safety, and effectiveness of outpatient operative hysteroscopy, with similar success rates and complication profiles compared to procedures performed in the operating room, although some studies reported higher levels of pain during outpatient procedures (1-3) . Furthermore, cost-effectiveness studies support outpatient procedures by highlighting reduced hospital resource utilization and shorter recovery times for patients (4-6).

The HOPE study aims to evaluate this practice locally at the Centre Hospitalier Intercommunal de Créteil. This prospective monocentric observational study will include approximately 400 patients over a two-year period (July 2025 - May 2027). The primary objective is to compare the success rates of operative hysteroscopies performed in the operating room versus those performed in an outpatient setting. Secondary objectives include assessment of perioperative and postoperative pain, patient satisfaction, complication rates, and the time to return to work.

Data will be collected from medical records and patient-reported outcomes using a satisfaction questionnaire. Inclusion of patients will follow the usual care pathway, without additional interventions or follow-up beyond standard clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥ 18 years

  -⁃ Undergoing operative hysteroscopy for intrauterine pathology
* Able to provid e informed non-opposition
* French-speaking

Exclusion Criteria:

* Patients with contraindications to hysteroscopy
* Pregnancy
* Inability to complete follow-up

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Adult women requiring operative hysteroscopy for intrauterine pathology
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
This will be assessed as an ordinal qualitative variable, with procedures classified into three categories:number of complete success, number of partial success, or number of failure. | The classification will be determined by the surgeon at the end of the procedure and documented in the operative report (baseline)

SECONDARY OUTCOMES:
Perioperative and postoperative pain Assessed using the Visual Analogue Scale (VAS) | During the procedure (if the patient is awake), immediately after the procedure, and at hospital discharge (baseline)
Patient satisfaction Assessed using a locally developed patient satisfaction questionnaire | At hospital discharge.(assessed up to 5 days)
Complications including uterine perforation, hemorrhage, and postoperative infection | Recorded during the procedure and immediately afterward (documented in the operative report and medical records), and up to 8 weeks postoperatively during the follow-up consultation if necessary.
4. Time to return to work Measured as the number of days of sick leave prescribed and actually taken. | Up to 8 weeks postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- CHI Créteil - Gynécologie et obstétrique, Créteil, France